CLINICAL TRIAL: NCT04942483
Title: Biomarkers in Preschool Children With Wheeze to TArget Therapy wIth inhaLed cORticosteroids (TAILOR): a Feasibility Study".
Brief Title: Using Tests in Preschool Children With Wheeze to Determine the Need for Inhaled Corticosteroid Therapy.
Acronym: TAILOR
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Collaborators: Asthma UK Centre for Applied Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: 21IC6984; 300524 (Registry Identifier: IRAS)
Record Dates: First submitted 2021-06-22; First posted 2021-06-28 (Actual); Results first posted 2025-04-11 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Wheezing
Keywords: Preschool; Wheeze; Wheezing; Inhaled Corticosteroids; ICS; Biomarkers
MeSH Terms: conditions — Respiratory Sounds | interventions — Fractional Exhaled Nitric Oxide Testing

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Preschool children with a history of wheeze, aged 1 to 5 years old: This is a pragmatic, observational study involving preschool children with wheeze aged one to five years old. All treatment and routine monitoring decisions will be at the discretion of their treating general practitioner (GP) or paediatrician (as per usual clinical practice), blinded to the study measurements.
  The following three biomarker tests will be performed a) atopic sensitisation, b) blood eosinophil count and c) FeNO (off-line method).
  Interventions: Diagnostic Test: Blood eosinophil count; Diagnostic Test: Atopic sensitization; Diagnostic Test: FeNO (offline method)

INTERVENTIONS:
Diagnostic Test: Blood eosinophil count — Peripheral blood eosinophil count will be measured from a finger prick blood sample, using the Haemocue machine, allowing a result in approximately 2 minutes. The test will allow to assess the presence or not of eosinophilia and if it can predict future wheezing exacerbations and response to inhaled corticosteroids (ICS).
Diagnostic Test: Atopic sensitization — Skin prick tests will be performed to: (a) house dust mite, (b) grass pollen, (c) tree pollen, (d) cat hair, (e) dog hair, as well as normal saline and histamine which will act as negative and positive controls respectively. In addition, skin prick tests will allow the assessment of which aeroallergen is the most useful predictor of outcomes in preschool children.
Diagnostic Test: FeNO (offline method) — The child will breathe normally into a sample bag that will be collected for later analysis of FeNO levels. The test will be performed twice.

SUMMARY:
Wheezing is common in preschool children and affects quality of life. Although asthma treatments such as inhaled steroids (ICS), which reduce swelling (inflammation) in the airways are used in this age group, they are often ineffective. That is because only some preschool children have the type of inflammation (known as Type 2 inflammation) that responds to ICS, thus many children are being unnecessarily exposed to side effects. It is difficult diagnosing Type 2 inflammation through history and examination, thus other indicators are needed to ensure ICS are only given to children who will benefit. These indicators are commonly known as biomarkers, and we are trying to find out if they are useful. We want to measure three biomarkers, without changing children's treatment. The first is blood eosinophils. which can be measured using a finger prick sample (like the blood drop used for measuring sugar levels in diabetic children). The second is to determine if allergic sensitization is present to allergens that are breathed in; these will be house dust mite, grass pollen, tree pollen, cat and dog hair. The final biomarker is a molecule that is produced in the airways of preschool children with Type 2 inflammation, called nitric oxide (NO). This is easily obtained, by having children breathe through a mask and collecting their breath in a bag, measuring NO later on. The children will be followed up with monthly electronic questionnaires and 3-monthly visits (virtual or face-to-face) for a year to evaluate whether these markers individually or in combination relate to subsequent wheezing outcomes, and how acceptable the measurements are to families using a questionnaire and focus group approach. The results will form the basis of the design of a national trial of biomarker-driven therapy in such children.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged one to five years old presenting to primary care or emergency department or urgent care centre or identified from primary care records and have been diagnosed with wheezing by their GP or paediatrician who has decided to prescribe any bronchodilator, ICS or montelukast on clinical grounds
2. Parents/Carers able to understand and familiarize themselves with the study and are willing to provide informed consent

Exclusion Criteria:

1. Inability to understand and cooperate with study procedures
2. Significant co-morbidity (respiratory or otherwise), for example cystic fibrosis (excluding atopic disorders such as eczema, allergic rhinitis and food allergy)
3. Withholding or withdrawal of informed consent
4. Severe procedural anxiety (needle phobia)
5. Child is already enrolled in another study involving investigational medicinal product (CTIMP)
6. History of anaphylaxis or near-fatal asthma that resulted in intubation / assisted ventilation.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children aged one to five years old presenting either to primary care with wheezing episodes or to emergency departments or urgent care centres with an acute attack of wheeze or children identified from primary care records and have been diagnosed with wheezing by their GP or paediatrician.
Sampling Method: Non-Probability Sample
Enrollment: 118 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Bush, MD FHEA FRCP FRCPCH FERS FAPSR, Principal Investigator — Imperial College London
Locations (1):
- John Radcliffe Hospital, Oxford, United Kingdom

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Only children 1-5 years old were considered enrolled. Their parents/guardians were not considered as enrolled. They signed the consent form for enrolment and complete the monthly questionnaires during follow-up on behalf of their child. No interventions were performed in this study. There were no arms in this study, only a single group followed in an identical manner.
Groups:
- Preschool Children Aged 1 to 5 Years Old: Preschool children with a history of ≥1 doctor-diagnosed acute wheeze attack of any severity, in the year prior to baseline measurement.
Period: Overall Study
Arm/Group | Preschool Children Aged 1 to 5 Years Old
Started | 118
Completed | 95
Not Completed | 23

BASELINE CHARACTERISTICS:
Population: Data on children's age, gender and ethnicity were provided by their parents. The baseline analyses apply only to preschool children aged 1-5 years old (not their parents).
Arm/Group | Preschool Children Aged 1 to 5 Years Old
Number analyzed (Participants) | 95
Age, Continuous [Median (Full Range); unit: months] | 35 [13 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 86
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 95
Blood eosinophil count [Median (Full Range); unit: cells/μL] | 400 [0 to 1400]
Fractional exhaled nitric oxide [Median (Full Range); unit: ppb] | 8 [0 to 18.5]
Atopy [Count of Participants; unit: Participants] | 45

OUTCOME MEASURES:

1. Primary Outcome: Wheeze Attacks
Description: Defined as requiring an unscheduled healthcare visit to the ED or GP.
Time Frame: 1-year follow-up
Population: Data only applies to children aged 1-5 years old. There were no arms in this study, only a single group followed in an identical manner.
Measure: Median (Full Range); unit: Wheeze attacks
Groups:
- Preschool Children Aged 1-5 Years: Preschool children aged 1-5 years followed for a period of 12 months. There were no arms in this study, only a single group followed in an identical manner.
Arm/Group | Preschool Children Aged 1-5 Years
Number analyzed (Participants) | 95
Wheeze attacks | 1 [0 to 9]

2. Secondary Outcome: Days Out of Nursery
Description: Children unable to attend childcare facility due to a wheeze attack. There were no arms in this study, only a single group followed in an identical manner.
Time Frame: 1 year follow-up period
Population: Data only applies to children aged 1-5 years old and not their parents. There were no arms in this study, only a single group followed in an identical manner.
Measure: Median (Full Range); unit: days
Groups:
- Preschool Children Aged 1-5 Years Old: Days out of nursery preschool children aged 1-5 years old needed to take due to a wheeze attack in the 12 month follow-up period.
Arm/Group | Preschool Children Aged 1-5 Years Old
Number analyzed (Participants) | 95
days | 3 [0 to 33]

3. Secondary Outcome: Parents Days Out of Work
Description: Days out of work parents needed to take because of their child's wheeze attack. There were no arms in this study, only a single group followed in an identical manner.
Time Frame: 1 year follow-up period
Population: Data only apply to parents of preschool children. There were no arms in this study, only a single group followed in an identical manner. Every month parents would be asked to state whether they needed to take any days of work due to their child's wheeze.
Measure: Median (Full Range); unit: days
Groups:
- Parents of Preschool Children: Days out of work parents of preschool children needed to take during the 12-month follow-up period because of their child's wheeze. There were no arms in this study, only a single group followed in an identical manner.
Arm/Group | Parents of Preschool Children
Number analyzed (Participants) | 95
days | 3 [0 to 33]

4. Other Pre Specified Outcome: Acceptability of Biomarker Tests by Parents
Description: The acceptability of the three biomarker tests by parents to be used in clinical practice was assessed through focus group discussions.
Time Frame: 12-months
Population: Only 16 out of 95 parents agreed to participate in these focus group discussions.
Measure: Count of Participants; unit: Participants
Groups:
- Parents of Preschool Children: Parents of preschool children with wheeze
Arm/Group | Parents of Preschool Children
Number analyzed (Participants) | 16
Participants | 16

ADVERSE EVENTS:
Time Frame: Only during biomarker testing (i.e., at single baseline visit and at second visit 3 months post-baseline)
Description: Adverse events were recorded for the biomarker measurements but not during the observation period.
Groups:
- Preschool Children Aged 1 to 5 Years Old: Adverse events were recorded for the biomarker measurements (i.e., at single baseline visit and at second visit 3 months post-baseline) but not during the observation period.
Arm/Group | Preschool Children Aged 1 to 5 Years Old
All-Cause Mortality (participants affected / at risk) | 0/95
Serious Adverse Events (participants affected / at risk) | 0/95
Other Adverse Events (participants affected / at risk) | 0/95

LIMITATIONS AND CAVEATS:
FeNO measurements were not obtained in all children due to delayed appreciation that the gas collection bag was faulty. However, a mitigation strategy was utilised to increase the number of children who had FeNO recorded. Children with FeNO measurement at baseline and those with a FeNO measurement in the second, but not baseline testing were combined, giving 68 children with FeNO measurements.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/83/NCT04942483/Prot_SAP_000.pdf